CLINICAL TRIAL: NCT06921226
Title: Intra-personal and Interpersonal Psychological Processes Involved in Risk-taking and Suicidal Behaviors Among Vulnerable Adolescents and Adults
Brief Title: Exploratory Analysis of Interpersonal and Intrapersonal Psychological Processes Implied in Risk-taking and Suicidal Behaviors, in Adult and Adolescent At-risk
Acronym: RISKY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Metropole Savoie (Other)
Collaborators: Centre Hospitalier Spécialisé de la Savoie (Chambéry) (Unknown); Université Savoie Mont Blanc (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CHMS24005
Record Dates: First submitted 2025-03-25; First posted 2025-04-10 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Suicidal Ideas; Suicidal Ideation; Risk-taking
Keywords: Risk-taking behaviors; Impulsivity; Interpersonal needs; Suicidal ruminations; Suicidal behaviors; BART
MeSH Terms: conditions — Suicidal Ideation; Risk-Taking; Impulsive Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Procedure based on questionnaires and a computer task (Experimental): This study begins with an initial screening phase. Only individuals exhibiting suicidal ideation and/or behavior, as identified by at least one affirmative response out of six on the C-SSRS scale (Posner et al., 2011), will be eligible to proceed with the study.
  Subsequently, they will complete seven questionnaires and one computer task:
  * Risk-taking behaviors via a computer task via the Balloon Analogue Risk Task (BART, Lejuez et al., 2002, 2007) and questionnaires (NRTB and PRTB, Duell et al., 2020; Fryts et al., 2024)
  * Decision-making styles (GDMS, Scott and Bruce, 1995)
  * Impulsivity (UPPS-Short, Billieux et al., 2012)
  * Depressive symptoms (CES-D, Fuhrer and Rouillon, 1989)
  * Interpersonal needs (INQ, Landrault et al., 2019)
  * Suicidal ruminations (SRS, Rogers et al., 2022)
  Interventions: Other: Psychological Processes; Other: Risk-taking variables; Other: Suicidal ideation and behavior

INTERVENTIONS:
Other: Psychological Processes — * The sense of thwarted belonging and perceived burden will be measured using the Interpersonal Needs Questionnaire (INQ; Van Orden et al., 2012). The back-translated French version by Landrault et al. (2019) will be used. This scale is based on a seven-point Likert scale, ranging from 1 (not at all true for me) to 7 (very true for me).
  * To assess impulsivity, we will use the short version of the UPPS validated in French by Billieux and colleagues (2012). It comprises 20 items divided into 5 dimensions (negative urgency, positive urgency, lack of premeditation, lack of perseverance and sensation seeking). Participants were asked to respond on a Likert scale from 1 ("I strongly agree") to 4 ("I strongly disagree").
  * We will use the French version of the SRS (Suicidal Rumination Scale, Rogers et al., 2022), back-translated for this study. This eight-item scale assesses suicidal ruminations.
Other: Risk-taking variables — * One of the behavioral tasks based on a real-life model of risky decision-making is BART (Lejuez et al., 2002, 2007). It is based on a conceptual framework of balance between reward and loss potential (Leigh, 1999; Lejuez et al., 2002).
  * We will measure one of the cognitive aspects of risk-taking behavior, especially the general cognitive decision-making styles (GDMS, from Scott and Bruce, 1995; Gerard et al., 2016).
  * We will measure negative (NRTB , Duell et al., 2020) and positive (PRTB, Fryts et al., 2024) self-reported risk-taking behaviour.
Other: Suicidal ideation and behavior — Suicidal ideation and behavior were measured using the screening grid, the Columbia Suicide Severity Rating Scale (C-SSRS screen version, Posner, Brown, Stanley et al., 2011). It is composed of 6 questions, which take into account the potential method of suicide, the presence of suicidal intent and/or ideation with a plan or intention. This scale has high reliability and validity in general paediatric emergencies (Scudder et al., 2023) and psychiatric samples (Campos et al., 2023).
  It classifies people as being at low or high risk of suicide, based on the presence or absence of significant active suicidal ideation in the last three months.

SUMMARY:
In a recent report, Santé Publique France (2023), reported that 4.2% of 18-85 year-olds had thought about suicide in the last 12 months, and 6.8% had attempted suicide in their lifetime and 0.5% in the last year. Even more recently, the DREES (Direction de la recherche, des études, de l'évaluation et des statistiques auprès des Ministères Sociaux) published a report on May 16, 2024, showing a sharp rise in hospitalization rates for self-inflicted acts among female patients aged between 10 and 24, with a peak around age 15. Two-thirds of these hospitalizations for self-inflicted injuries are related to deliberate drug intoxication. Depression, bipolar disorders and schizophrenia spectrum disorders (among other psychological disorders) are known risk factors for suicide, which is the leading cause of death in this clinical context. In addition to these formalized psychopathological elements, risk behaviors underpinned by psychological processes common to suicide attempts are suspected and need to be studied in depth.

Research into psychiatry and the psychopathology of suicide has identified a number of risk and protective factors. These psychological determinants - or processes - act alongside other key factors such as the environment and social ties. Life contexts can have an impact on health, and more specifically on the psychopathology of individuals, through disturbances of a biological, psychological and social nature. It is important to be able to describe what processes are at work and how they explain the development and maintenance of behaviours that put one's life and health at risk. This is part of a preventive approach to mental health. We suggest that the study of psychological processes such as suicidal ruminations, impulsivity and interpersonal needs (e.g. the interpersonal theory of suicide) is necessary to understand their involvement in risk-taking and suicidal behavior. To our knowledge, few studies of this type are underway in France, particularly with vulnerable clinical populations (adolescents/adults). The inclusion of a process-centered approach (Kinderman, 2015), in a transdiagnostic and preventive way, constitutes an innovative approach.

DETAILED DESCRIPTION:
The aim of this study is to describe psychological processes that contribute to risk-taking and suicidal behaviors.

The primary objective of this study is: To examine the fit of an Structural Equation Model (SEM) of risk-taking and suicidal behaviors and ideation, and explain those self-destructive behavior can possibly affected by Perceived Burdensomeness (PB) and Thwarted Belongingness (TB), Impulsivity and Suicidal Ruminations (SR) among with suicidal ideations.

This study will address the following secondary objectives:

1. To explore the mediating effect of risk-taking, as a behavioral variable, on the relationship between suicidal ideation and behavior and impulsivity.
2. To explore the mediating effect of risk-taking, as a self-reported variable, on the relationship between suicidal ideation and behavior and impulsivity.
3. To explore the mediating effect of risk-taking, as a cognitive variable, on the relationship between suicidal ideation and behavior and impulsivity.
4. To explore the mediating effect of PB on the relationship between SR and suicidal ideation and behavior.
5. To explore the mediating effect of TW, on the relationship between SR and suicidal ideation and behavior.
6. To explore the mediating effect of SR on the relationship between suicidal ideation and behavior and impulsivity.

The effect of developmental status (adult versus adolescent), will be considerated as a co-variate.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-65 years
* Adolescent population considered as at risk in mental health : admitted to the peadiatric department (CHMS).

or - Adult population : user of the Espoir73 association (an association for adults with a mental health problem) or users of SM@RT (CHS, a psycho-social rehabilitation center for adults with a mental illness).

Exclusion Criteria:

- No suicidal ideation or behaviors (none " Yes " response at the 6 questions of the C-SSRS screen version).

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Suicidal ideation and behaviors | At inclusion
  C-SSRS score (screen version) out of 6

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CH Métropole Savoie, Chambéry, Savoie
  - Centre Hospitalier Spécialisé de la Savoie (CHS), Bassens
  - ESPOIR73, Francin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McHugh CM, Chun Lee RS, Hermens DF, Corderoy A, Large M, Hickie IB. Impulsivity in the self-harm and suicidal behavior of young people: A systematic review and meta-analysis. J Psychiatr Res. 2019 Sep;116:51-60. doi: 10.1016/j.jpsychires.2019.05.012. Epub 2019 May 17. PMID 31195164
- [Background] Rogers ML, Gallyer AJ, Joiner TE. The relationship between suicide-specific rumination and suicidal intent above and beyond suicidal ideation and other suicide risk factors: A multilevel modeling approach. J Psychiatr Res. 2021 May;137:506-513. doi: 10.1016/j.jpsychires.2021.03.031. Epub 2021 Mar 26. PMID 33812323
- [Background] Sastre-Buades A, Alacreu-Crespo A, Courtet P, Baca-Garcia E, Barrigon ML. Decision-making in suicidal behavior: A systematic review and meta-analysis. Neurosci Biobehav Rev. 2021 Dec;131:642-662. doi: 10.1016/j.neubiorev.2021.10.005. Epub 2021 Oct 5. PMID 34619171
- [Background] Tomova, L., Andrews, J. L., & Blakemore, S.-J. (2021). The importance of belonging and the avoidance of social risk taking in adolescence. Developmental Review, 61, 100981. https://doi.org/10.1016/j.dr.2021.100981
- [Background] Tucker RP, Hagan CR, Hill RM, Slish ML, Bagge CL, Joiner TE Jr, Wingate LR. Empirical extension of the interpersonal theory of suicide: Investigating the role of interpersonal hopelessness. Psychiatry Res. 2018 Jan;259:427-432. doi: 10.1016/j.psychres.2017.11.005. Epub 2017 Nov 6. PMID 29128621
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671